CLINICAL TRIAL: NCT02090894
Title: Effect of Dermal Rejuvenation on the UVB Response of Geriatric Skin
Acronym: Laser Genesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ally-Khan Somani, M.D., Ph.D., Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1105005442
Record Dates: First submitted 2014-01-28; First posted 2014-03-18 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-05

CONDITIONS: Pre-cancerous Geriatric Skin

ARMS (1):
- UV Light (Experimental)
  Interventions: Device: UV Light (Laser Genesis)

INTERVENTIONS:
Device: UV Light (Laser Genesis)

SUMMARY:
The objective of this study is to examine the ability of dermal rejuvenation therapies to protect geriatric skin from ultraviolet light (UVB)-induced carcinogenesis. Skin cancers (including basal cell carcinoma and squamous cell carcinoma) are the most common types of malignancy and are related to UVB exposure in sunlight. UVB-irradiation of skin causes specific DNA damage to keratinocytes that can lead to cancer-causing mutations if they are allowed to persist in proliferating cells. Moreover, the incidence of skin cancers is much greater in elderly over younger individuals. The objective of the present study is to build upon our previous data and test the effect of a non ablative Nd:YAG laser (LaserGenesis) of a localized area of skin on dermal IGF-1 production and UVB-mediated keratinocyte effects. Treatment of skin using a non ablative high-peak power microsecond pulsed 1064 nm Nd:YAG laser (Cutera's LaserGenesisTM laser) leads to papillary dermal heating. The laser targets the microvasculature and stimulates collagen production while protecting the epidermis. Generally, Laser Genesis is used clinically to improve irregularities in the contour, texture, and color of the skin. Laser Genesis is also used to help treat photoaging by increasing collagen formation, suggesting that it stimulates fibroblast activity and thus possibly increases levels of protective IGF-1.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects older than 65 years will be enrolled.
* Subject's skin type must be "Fair", Fitzpatrick type I or II.

Exclusion Criteria:

* Subjects who have underlying diseases that could affect wound healing (eg, diabetes mellitus)
* on medications that are known photosensitizers,
* or have a history of abnormal scarring (eg, keloids) will be excluded.

Subjects will be asked the screening questions below as part of the inclusion/exclusion criteria

* How old are you?
* Do you regularly use tanning beds?
* Are you being treated with light therapy?
* Have you had any diseases that got worse when you went in the sun?
* Are you taking any medications that warn you to stay out of the sun?
* Have you ever had a reaction to medications that were applied to your skin?
* When cuts or wounds on your skin heal, are the scars abnormally large or take a long time to heal?
* Do you have diabetes mellitus or have you ever had high blood sugar?

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Department of Dermatology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- UV Light: UV Light (Laser Genesis). 1064 nm laser at a fluence of 13-16 J/cm2 and a pulse width of 0.3 ms and a 5 mm spot size
Period: Overall Study
Arm/Group | UV Light
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- LaserGenesis Treatment: 1064 nm laser at a fluence of 13-16 J/cm2 and a pulse width of 0.3 ms and a 5 mm spot size
Arm/Group | LaserGenesis Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Difference in Basal Layer Keratinocytes Positive for Both Ki67 and Thymine Dimers
Description: Number of double positive cells per 1000 total basal layer keratinocytes
Time Frame: untreated and LaserGenesis treated, three months after treatment, 24 hours after 350 J/m2 of UVB
Population: untreated and laser treated biopsies were taken from each subject
Measure: Mean (Standard Deviation); unit: positive cells/1000 basal layer cells
Arm/Group | LaserGenesis Treatment
Number analyzed (Participants) | 11
positive cells/1000 basal layer cells
  Untreated skin | 21.5 (16.3)
  Laser-treated skin | 14.7 (13.4)

2. Secondary Outcome: Relative Level of IGF-1 mRNA in the Skin
Description: IGF-1 mRNA per 100,000 beta-2 microglobulin mRNA. Beta-2 microglobulin mRNA was used as a reference gene for this assessment and that the data represent number of copies IGF-1/100,000 copies b2-microglobulin.
Time Frame: untreated and LaserGenesis treated, three months after treatment
Population: untreated and laser treated biopsies were taken from each subject
Measure: Mean (Standard Error); unit: relative mRNA
Arm/Group | LaserGenesis Treatment
Number analyzed (Participants) | 11
relative mRNA
  Untreated skin | 70.5 (22.1)
  Laser-treated skin | 115.1 (43.9)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- LaserGenesis Treatment: 1064 nm laser at a fluence of 13-16 J/cm2 and a pulse width of 0.3 ms with a 5 mm spot size
Arm/Group | LaserGenesis Treatment
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No